CLINICAL TRIAL: NCT05295524
Title: Description of the Short-term Effects of KAFTRIO® by Continuous Monitoring With the PHEAL-CR-K Application in Real Life in Patients With Cystic Fibrosis Eligible for KAFTRIO® Treatment
Acronym: PHEAL-KAFTRIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021_0201
Record Dates: First submitted 2022-02-18; First posted 2022-03-25 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: prospective, open-label, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Cystic Fibrosis, with KAFTRIO® treatment prescription (Experimental): Patients with Cystic Fibrosis, for whom treatment with KAFTRIO® is prescribed, regardless of previously prescribed CFTR modulator treatments.
  Interventions: Other: Kaftrio utilization in real life

INTERVENTIONS:
Other: Kaftrio utilization in real life — daily utilization of PHEAL-CR-K application at home and VOC (volatile organic compound) measure of exhaled air for a group of the patients

SUMMARY:
This is a prospective, open-label, multicenter study (1 year) with 50 patients with cystic fibrosis for whom treatment with KAFTRIO® is prescribed.Cystic fibrosis is a rare autosomal recessive hereditary disease linked to a mutation of the CFTR (Cystic Fibrosis Transmembrane Regulator) protein gene. For the majority of patients, no treatment with a CFTR protein modulator was available until the arrival of the KAFTRIO® triple therapy (ivacaftor/tezacaftor/elexacaftor). Clinical studies on this triple therapy demonstrate significant improvements in FEV (forced vital capacity) and also very rapid health improvement of patients. However, there is a lack of data recorded in real life at home by patients to trace the evolution curves of health parameters and patient perceptions from the first days after initiation of treatment. The PHEAL-CR-K application, specially developed for the study, makes it possible to collect physiological parameters and perceptions collected via connected objects or declared manually in the application. These data will reflect the evolution of the parameters from the start of the treatment and over a period of 3 months. In addition, the composition of volatile organic compounds (VOCs) of the air exhaled in the early phase of treatment with KAFTRIO® will be monitored for the group of patients followed at Foch Hospital. Exhaled air is an ideal biological fluid for clinical monitoring (non-invasive collection and real-time analysis). In cystic fibrosis, biomarkers in the exhaled air have been correlated with functional and clinical parameters. The objective is to collect the air exhaled before initiating treatment with KAFTRIO® and during treatment, to identify VOCs whose expression would be modified early. Changes in the composition of the exhaled air will be correlated with follow-up clinical data collected with the PHEAL-CR-K application and with functional data obtained during measurements of breath by spirometry (FEV) and sweat concentrations of chloride ions collected at the during a sweat test. The identified COVs could become early predictive biomarkers of clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patients with Cystic Fibrosis eligible for KAFTRIO®
* Patients for which KAFTRIO® treatment is prescribed, including patients previously treated with other CFTR modulators (ORKAMBI®, KALYDECO®, SYMKEVI®)
* Patients who signed the informed consent form
* Patients affiliated to a health insurance plan
* Patients equipped with a smartphone and having a Wifi connection at home

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient who does not speak or understand French
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Collection of the different remarkable events declared in the application (adverse events and favorable events measured by perception scales) | 1 year
  Collection of the different remarkable events declared in the application (adverse events and favorable events) between Day 0 and Day 60 +/-30 days
  A great number of data will be collected from the indications declared by the patient at home and cannot be summarized in the title.
  The originality of the study is the collection in real life facilitated by the provision of connected objects and the functionnalities of the PHEAL-CR-K application

SECONDARY OUTCOMES:
FEV1 (Forced Expiratory Volume in one second) measurements by portable spirometer at Day 0 and Day 60 +/-30 days, between the consultation before introduction of the drug and the first follow-up visit | 1 year
Daily evolution or over the course of the measurements carried out during the follow-up period of FEV1 (Forced Expiratory Volume in one second) with a spirometer | 1 year
  The patient performs the measurements at home with a connected spirometer allowing to inform the respiratory capacity through the measurement of FEV1
Daily evolution or over the course of the measurements carried out during the follow-up period of weight (in kilograms) and body mass index (in kg/m^2) | 1 year
  The patient has a connected balance at home to measure his weight. The body mass index is calculated by the application, with the height (in meters) indicated by the patient
Daily evolution or over the course of the measurements carried out during the follow-up period of oxygen saturation collected by a connected watch | 1 year
  The patient wears a connected watch on day that measures the oxygen saturation in blood and reports the data in the application
Daily evolution or over the course of the measurements carried out during the follow-up period of heart rate and respiratory rate measured by connected watch and mattress pad | 1 year
  The heart rate is measured at home by a connected watch (on day). A connected mattress pad measures the heart rate and respiratory rate at rest (during the sleep).
Evolution of respiratory exacerbations by the declaration in the application of clinical perceptions (surveys to describe the cough and the expectoration) and/or declaration of antibiotic prescription | 1 year
  Respiratory exacerbations are declared at home by the patient in the application :
  * Surveys allow to describe the cough (frequency, type, moment) and the expectorations (clinical perception)
  * A feature is present to declare antibiotic prescription
Collection of reported perceptions (cough, sputum, nasal secretions, dyspnea, fatigue, sleep dyspnea, sleep, appetite, other) via visual analog scales (from zero to 4, from the better to the worse outcome) | 1 year
  A list of perceptions are reported in the application (cough, sputum, nasal secretions, dyspnea, fatigue, sleep dyspnea, sleep, appetite, other), with scales.
  The patient declares the perceptions at home, daily or over the course of the study, by using the 3 scales for each indicator. The final score is the mean of the 3 scales. The minimum value is 0, the maximum value is 4. The highest score means a worse outcome.
Collection of KAFTRIO® compliance (missed medication) | 1 year
Collection of anciliary antibiotic therapies and care provided (declaration in the application) | 1 year
  The patient can declare in the application the prescription of anciliary antibiotic therapies and care provided. This is not a measure but an complementary information of the patient health.
Assessment of the Cystic Fibrosis Questionnaire-Revised (CFQ-R) score (scale 0-100, with higher score indicating better health-related quality of life) before/after (at Day1 at inclusion and at Day 60+/-30 at the end of the study) | 1 year
Evaluation of VOC (volatil organic compound) profiles in exhaled air at ay D0 and variation of these profiles after treatment (during the first week and Day 60 +/-30 days) | 1 year
Identification of VOCs (volatil organic compound) whose abundance is modified by the KAFTRIO® treatment | 1 year
Correlation of VOC (volatil organic compound) changes to clinical and paraclinical efficacy data: remarkable events, reported events, reported perceptions, FEV1 (Forced Expiratory Volume in one second), sweat chloride ion concentration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Grenet, Principal Investigator — Foch Hospital
Locations (1):
- Grenet Dominique, Suresnes, France

IPD SHARING:
Plan to Share IPD: Undecided